CLINICAL TRIAL: NCT06398288
Title: Adjunctive Use of Dermal Matrix to Compensate Dimensional Changes in the Reconstructive Therapy of Peri-implantitis: Multi-Center Randomized Controlled Trial
Brief Title: Adjunctive Use of Dermal Matrix to Compensate Dimensional Changes in the Reconstructive Therapy of Peri-implantitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18002604
Record Dates: First submitted 2024-04-27; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Oracell group) (Experimental): Mechanical detoxification using curettes + NiTi brushes + EA (GalvoSurge) for 2 minutes + a mixture of anorganic bovine bone (Straumann Xenograft, Straumann) and cortical mineralized/demineralized allograft (Oragraft, Lifenet Health) + dermal matrix on the buccal aspect (Oracell, Lifenet Health)
  Interventions: Other: Dermal matrix (Oracell, LifeNet, USA)
- Control group (no Oracell group) (Experimental): Control group: Mechanical detoxification using curettes + NiTi brushes + EA (GalvoSurge) for 2 minutes + a mixture of anorganic bovine bone (Straumann Xenograft, Straumann) and cortical mineralized/demineralized allograft (Oragraft, Lifenet Health)
  Interventions: Other: No dermal matrix

INTERVENTIONS:
Other: Dermal matrix (Oracell, LifeNet, USA) — Mechanical detoxification using curettes + NiTi brushes + EA (GalvoSurge) for 2 minutes + a mixture of anorganic bovine bone (Straumann Xenograft, Straumann) and cortical mineralized/demineralized allograft (Oragraft, Lifenet Health) + dermal matrix on the buccal aspect (Oracell, Lifenet Health)
  Arms: Test group (Oracell group)
Other: No dermal matrix — Mechanical detoxification using curettes + NiTi brushes + EA (GalvoSurge) for 2 minutes + a mixture of anorganic bovine bone (Straumann Xenograft, Straumann) and cortical mineralized/demineralized allograft (Oragraft, Lifenet Health)
  Arms: Control group (no Oracell group)

SUMMARY:
One critical element regarded to successfully resolve peri-implantitis is to efficiently decontaminate the contaminated implant surface. Mechanical, pharmacological and chemical strategies have been proposed to eliminate bacterial plaque and remnants from the implant surface. However, evidence has not demonstrated superiority of a given detoxification agent/strategy. Recently, the electrolytic approach has been indicated for the surgical detoxification in the management of peri-implantitis. For the electrolytic approach (EA) the implant has to be loaded negatively with a voltage and a maximum current of 600 mA. This is achieved by a device (GS1000, GalvoSurge Dental AG, Widnau, Switzerland) providing the voltage and pumping a sodium formiate solution through a spray-head, which has to be pressed into the implant by finger pressure to achieve an electrical contact.

Another critical aspect in the management of peri-implantitis is related to the esthetic sequelae associated with disease resolution. Sanz-Martin et al. in a systematic review demonstrated that reconstructive therapy is less prone to exhibit mucosal recession when compared to resective therapy. Nonetheless, it seems to be unavoidable no matter the surgical intervention. Aiming at attenuating these changes, Schwarz et al. noted that the adjunctive use of connective tissue grafts may enhance the height of the mucosal level, which in turn may impact upon the esthetic outcome. Therefore, the research question is the following: What is the clinical, radiographic and 3D volumetric effectiveness of dermal matrix to improve the outcome of reconstructive therapy of peri-implantitis-related bone defects? The study is to be performed in two centers: Center of Implantology, Oral and Maxillofacial in Badajoz (Spain) and Clinical PerioCentrum Ortiz-Vigon in Bilbao (Spain)

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with peri-implantitis-related intrabony defects
* All subjects had dental implants with screw-retained or cement-retained fixed or removable implant-supported prosthesis for a minimum of 36 months.
* All patients in age of 18 to 80, non-smokers
* With no presence of systemic disease or medication known to alter bone metabolism, and partial or complete edentulous patients that have no active periodontal disease.

Exclusion criteria:

* Peri-implantitis-related supra-crystal or combined defects
* Pregnancy or lactation
* History of or current smokers
* Uncontrolled medical conditions,
* Cement-retained restorations,
* Lacking keratinized mucosa (≤2mm) on the lingual or buccal implant sites.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of disease resolution of peri-implantitis (%) | 12 months
  No bleeding, no pocket depth ≥6mm, no progressive bone loss. Appraised in %

SECONDARY OUTCOMES:
Reduction in mm of mucosal recession | 12 months
  Migration of the mucosal margin from baseline position in relation to the implant-abutment/prosthesis connection. Appraised in mm
Evolution of microbial profile (characteristics of the microbiota) | 12 months
  Microbiological samples will be taken with sterile endodontic paper points (Absorbent paper point size 30, Denstsply, Maillefer, Ballaigues, Switzerland) from the peri-implant sulcus of patients with implants diagnosed with peri-implantitis. In the event that the same patient has several implants with a diagnosis of peri-implantitis, separate samples will be taken from each peri-implant environment.
  * T=0. Submucosal microbiological sampling prior to the non-surgical phase. Before instrumentation. Intact environment.
  * T=1. Submucosal microbiological sampling prior to the surgical phase. Before the start of surgery. Environment evolved after instrumentation.
  * T=2. Submucosal microbiological sampling after 2 weeks of reconstructive surgery. After removing sutures, perform sampling.
  * T=3. Submucosal microbiological sampling 6 months of follow-up.
  * T=4. Submucosal microbiological sampling 12 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Monje, DDS, Principal Investigator — Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxiofacial, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Regidor E, Ortiz-Vigon A, Romandini M, Dionigi C, Derks J, Sanz M. The adjunctive effect of a resorbable membrane to a xenogeneic bone replacement graft in the reconstructive surgical therapy of peri-implantitis: A randomized clinical trial. J Clin Periodontol. 2023 Jun;50(6):765-783. doi: 10.1111/jcpe.13796. Epub 2023 Mar 6. PMID 36802084
- [Result] Monje A, Pons R, Vilarrasa J, Nart J, Wang HL. Significance of barrier membrane on the reconstructive therapy of peri-implantitis: A randomized controlled trial. J Periodontol. 2023 Mar;94(3):323-335. doi: 10.1002/JPER.22-0511. Epub 2022 Dec 12. PMID 36399349